CLINICAL TRIAL: NCT05107128
Title: A Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Effect of SAGE-718 on Cognitive Function in Participants With Huntington's Disease
Brief Title: A Study to Evaluate the Effect of SAGE-718 on Cognitive Function in Participants With Huntington's Disease (HD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 718-CIH-201; 2021-005577-16 (EudraCT Number)
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive SAGE-718-matching placebo, orally, once daily (QD) for up to Day 84.
  Interventions: Drug: Placebo
- SAGE-718 (Experimental): Participants will receive SAGE-718, 1.2 milligrams (mg), capsules, orally, QD for Days 1 to 27, followed by 0.9 mg for the remainder of the treatment period up to Day 84.
  Interventions: Drug: SAGE-718

INTERVENTIONS:
Drug: SAGE-718 — Oral capsules.
  Arms: SAGE-718
Drug: Placebo — SAGE-718-matching oral capsules.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the effect of SAGE-718 on cognitive performance and functioning in participants with HD.

ELIGIBILITY:
Inclusion Criteria:

1. Meet all the following criteria for HD at Screening (Days -28 to -2):

   1. Genetically confirmed disease with huntingtin gene CAG expansion greater than or equal to (≥) 36.
   2. At screening, Unified Huntington's Disease Rating Scale (UHDRS)-Total Functional Capacity (TFC) score greater than (>) 6 and less than (<)13, suggesting no more than a moderate level of functional impairment.
   3. No features of juvenile HD.
2. Score of 15 to 25 (inclusive) on the Montreal Cognitive Assessment (MoCA) at screening indicating the presence of cognitive impairment.
3. Be willing to invite a study partner, if available, who is reliable, competent, and at least 18 years of age to participate in the study.
4. Be ambulatory (use of assistance devices such as a walker or cane is acceptable, as is occasional use of wheelchair, as judged by the investigator. Individuals requiring a wheelchair on a regular basis are excluded), able to travel to the study center, and, as judged by the investigator, is likely to be able to continue to travel to the study center to complete study visits for the duration of the study.
5. Completion of Huntington's Disease Cognitive Assessment Battery (HD-CAB) Trail Making-B Test in less than 240 seconds at Screening (Days -28 to -2).

Exclusion Criteria:

1. Have participated in a previous clinical study of SAGE-718, have previous exposure to gene therapy, have participated in any HD investigational drug, biologic, or device trial within 180 days, or a non-HD drug, biologic, or device trial within 30 days or 5 half-lives (whichever is longer).

   (Note: Participants with confirmation of enrollment in the placebo arm of these trials would not be excluded.)
2. Have a diagnosis of an ongoing neurodegenerative condition other than HD, including but not limited to Alzheimer's Disease, vascular dementia, dementia with Lewy bodies, or Parkinson's Disease.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-10-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (46):
- United States (31):
  - Sage Investigational Site, Little Rock, Arkansas
  - Sage Investigational Site, La Jolla, California
  - Sage Investigational Site, Los Angeles, California
  - Sage Investigational Site, Sacramento, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Washington D.C., District of Columbia
  - Sage Investigational Site, Boca Raton, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Honolulu, Hawaii
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Indianapolis, Indiana
  - Sage Investigational Site, Iowa City, Iowa
  - Sage Investigational Site, Kansas City, Kansas
  - Sage Investigational Site, Baltimore, Maryland
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Farmington Hills, Michigan
  - Sage Investigational Site, Buffalo, New York
  - Sage Investigational Site, New York, New York
  - Sage Investigational Site, Chapel Hill, North Carolina
  - Sage Investigational Site, Durham, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Toledo, Ohio
  - Sage Investigational Site, Philadelphia, Pennsylvania
  - Sage Investigational Site, Charleston, South Carolina
  - Sage Investigational Site, Memphis, Tennessee
  - Sage Investigational Site, Nashville, Tennessee
  - Sage Investigational Site, Houston, Texas
  - Sage Investigational Site, Richmond, Virginia
  - Sage Investigational Site, Kirkland, Washington
  - Sage Investigational Site, Spokane, Washington
  - Sage Investigational Site, Madison, Wisconsin
- Australia (4):
  - Sage Investigational Site, Westmead, New South Wales
  - Sage Investigational Site, Herston, Queensland
  - Sage Investigational Site, Bethlehem, Victoria
  - Sage Investigational Site, Nedlands, Western Australia
- Canada (3):
  - Sage Investigational Site, Halifax, Nova Scotia
  - Sage Investigational Site, North York, Ontario
  - Sage Investigational Site, Montreal, Quebec
- United Kingdom (8):
  - Sage Investigational Site, Tooting, London
  - Sage Investigational Site, Aberdeen
  - Sage Investigational Site, Birmingham
  - Sage Investigational Site, Cardiff
  - Sage Investigational Site, Leeds
  - Sage Investigational Site, Newcastle upon Tyne
  - Sage Investigational Site, Plymouth
  - Sage Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at investigative sites from 26 January 2022 to 03 October 2024.
Pre-assignment Details: A total of 309 participants with Huntington's disease (HD) were screened, of which 189 participants were randomized to receive either SAGE-718 or placebo.
Groups:
- Placebo: Participants received SAGE-718-matching placebo, orally, once daily (QD) for up to Day 84.
- SAGE-718: Participants received SAGE-718, 1.2 milligrams (mg), capsules, orally, QD for Days 1 to 27, followed by 0.9 mg for the remainder of the treatment period up to Day 84.
Period: Overall Study
Arm/Group | Placebo | SAGE-718
Started | 94 | 95
Completed | 87 | 91
Not Completed | 7 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Withdrawal of Consent | 0 | 1
Not completed — Reason Not Specified | 2 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who initiated investigational product (IP) and had baseline and at least 1 post-baseline efficacy evaluation.
Groups:
- Placebo: Participants received SAGE-718-matching placebo, orally, QD for up to Day 84.
- SAGE-718: Participants received SAGE-718, 1.2 mg, capsules, orally, QD for Days 1 to 27, followed by 0.9 mg for the remainder of the treatment period up to Day 84.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAGE-718 | Total
Number analyzed (Participants) | 94 | 95 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (8.71) | 50.0 (9.07) | 51.1 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 40 | 88
  Male | 46 | 55 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 87 | 86 | 173
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 90 | 87 | 177
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 2 | 4
Symbol Digit Modalities Test (SDMT) Score [Mean (Standard Deviation); unit: score on a scale] — The SDMT evaluates the tracking of cognitive function over time and for the early detection of cognitive impairment. The test assesses sustained attention, processing speed, visual scanning, and psychomotor speed, with the total score reflecting the number of correct pairings (out of 110 possible) completed within 90 seconds. Scores range from 0 to 110, with higher scores indicating better cognitive performance.
  score on a scale | 27.9 (11.86) | 28.3 (11.24) | 28.1 (11.52)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the SDMT
Description: The SDMT evaluates the tracking of cognitive function over time and for the early detection of cognitive impairment. The test assesses sustained attention, processing speed, visual scanning, and psychomotor speed, with the total score reflecting the number of correct pairings (out of 110 possible) completed within 90 seconds. Scores range from 0 to 110, with higher scores indicating better cognitive performance.
Time Frame: Baseline, Day 84
Population: The FAS included all participants who initiated IP and had baseline and at least 1 post-baseline efficacy evaluation. The overall number of participants analyzed indicates the number of participants with data available for this analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 90 | 93
score on a scale | 2.0 (0.58) | 0.8 (0.57)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.1675, MMRM — The p-value was obtained from Mixed Model for Repeated Measures (MMRM) model which includes treatment, visit, treatment-by-visit interaction as categorical covariates, and SDMT score at baseline as a continuous covariate; Difference in Least Square (LS) Means = -1.1, 95% CI 2-sided [-2.7 to 0.5], Standard Error of Mean 0.81 — Difference was calculated as SAGE-718 - placebo

2. Secondary Outcome: Change From Baseline in the Unified Huntington's Disease Rating Scale (UHDRS) - Independence Scale
Description: The UHDRS is a multi-domain clinical rating scale for assessment of functional capacity in HD. Independence Scale, Part V of the UHDRS, is a single-item measure to assess a participant's ability to function independently in daily activities across all stages of HD. Total score ranges from 10 to 100, with higher scores indicating better functioning. Negative change from baseline indicates worsening in functional ability.
Time Frame: Baseline, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 91 | 93
score on a scale | -0.8 (0.64) | -1.5 (0.63)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.4872, MMRM — The p-value was obtained from MMRM model which includes treatment, visit, treatment-by-visit interaction as categorical covariates, and UHDRS - Independence Scale at baseline as a continuous covariate; Difference in LS Means = -0.6, 95% CI 2-sided [-2.4 to 1.1], Standard Error of Mean 0.90 — Difference was calculated as SAGE-718 - placebo

3. Secondary Outcome: Change From Baseline in the Trail Making Test Part B
Description: The Trail Making test is a speeded graphomotor test of visual attention and task switching. Part B includes a set-switching component that requires participants to connect a series of alternating numbers and letters in order from lowest to highest (i.e., 1-A-2-B-3-C) in the shortest time possible. The time limit to complete the task is 240 seconds, at which point the test is stopped and scored using the maximum allowable time if not yet completed. Greater time indicates greater impairment. Negative change from baseline indicates less impairment.
Time Frame: Baseline, Day 84
Population: Participants in the FAS who completed the Trail Making Test Part B at baseline within the allowable time limit (240 seconds) were included in this analysis. Participants who exceeded the 240-second limit at baseline were excluded. The overall number of participants analyzed reflects those with baseline results within the allowable time limit and at least one post-baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 65 | 75
seconds | -5.7 (4.41) | -10.7 (4.11)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.4089, MMRM — The p-value was obtained from MMRM model which includes treatment, visit, treatment-by-visit interaction as categorical covariates, and SDMT score at baseline as a continuous covariate; Difference in LS Means = -5.0, 95% CI 2-sided [-17.0 to 6.9], Standard Error of Mean 6.04 — Difference was calculated as SAGE-718 - placebo

4. Secondary Outcome: Change From Baseline in the One Touch Stockings of Cambridge (OTS-Mean Latency Until Correct Response)
Description: The OTS is a computerized test of executive function to assess problem-solving and planning ability. In this task, participants are shown a set of colored balls and must determine the minimum number of moves required to match a target arrangement by moving one ball at a time into one of two available locations. The goal is to perform the task using the smallest number of moves possible. The participant selects the correct number of moves from the options shown on the screen. The time to correct response is measured. Longer times indicate greater impairment. Negative change from baseline indicates an improvement in performance.
Time Frame: Baseline, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 89 | 93
seconds | -4.56 (0.90) | -3.85 (0.88)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.5766, MMRM — The p-value was obtained from MMRM model which includes treatment, visit, treatment-by-visit interaction as categorical covariates, and a baseline value as a continuous covariate; Difference in LS Means = 0.70, 95% CI 2-sided [-1.78 to 3.19], Standard Error of Mean 1.26 — Difference was calculated as SAGE-718 - placebo

5. Secondary Outcome: Change From Baseline in the Paced Tapping Test (PTAP)
Description: The PTAP is a test of motor timing in which participants synchronize their finger taps with auditory pacing tones during an initial paced phase. This is followed by a self-paced phase, where the tones are removed, and the participant continues tapping until a final auditory cue signals the end of the test. The primary outcome is paced tapping consistency, calculated as the inverse of the standard deviation of the intertap intervals per millisecond (1/msec), with no range specified. Higher values indicate greater timing accuracy.
Time Frame: Baseline, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: 1/msec
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 90 | 92
1/msec | 0.710 (0.4552) | -0.157 (0.4510)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.1777, MMRM — The p-value was obtained from MMRM model which includes treatment, visit, treatment-by-visit interaction as categorical covariates, and baseline value as a continuous covariate; Difference in LS Means = -0.86, 95% CI 2-sided [-2.13 to 0.39], Standard Error of Mean 0.64 — Difference was calculated as SAGE-718 - placebo

6. Secondary Outcome: Change From Baseline in the Huntington's Disease Everyday Functioning (Hi-DEF) Home Subdomain Score
Description: Hi-DEF Scale: self-reported measure to capture difficulties experienced in daily life due to HD across 4 areas of functioning: At home, At work, Driving, & Relationships. Full scale comprises 40 items which ask participants to rate their functioning difficulty using 5-point Likert scale from 1 (No Difficulty) to 5 (Cannot do this anymore) on first 3 domains (home, work & driving), & 4-point scale from 1 (Never) to 4 (Always)for Relationships. Hi-DEF total score ranges from 0-154, higher score=greater difficulty. For Home subdomain, before scores can be calculated, data from item responses should be rescored so as: lowest item-level score=0 & highest item-level score= 4. Hence, Home subdomain has 15 items scored on 5-point Likert scale, 0 indicating no difficulty & 4 indicating cannot be done anymore, where total raw score of 0-60 are transformed to 0-100. Higher score=greater difficulty. Negative change from baseline=improvement in daily functioning.
Time Frame: Baseline, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 86 | 92
score on a scale | -4.6 (1.26) | -0.7 (1.23)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.0291, MMRM — The p-value was obtained from MMRM model which includes treatment, visit, treatment-by-visit interaction as categorical covariates, and Hi-DEF at baseline as a continuous covariate; Difference in LS Means = 3.9, 95% CI 2-sided [0.4 to 7.3], Standard Error of Mean 1.76 — Difference was calculated as SAGE-718 - placebo

7. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity (CGI-S) Cognitive Status Subdomain Score
Description: The CGI-S scale is a validated instrument developed by the National Institute of Mental Health specifically for use in clinical studies. Cognitive Status Subdomain is one of clinical global impression severity scales domains, for which clinicians generate ratings of the severity of the participant's condition over the past 7 days (including the day of the clinic visit). The responses are scored on a scale ranging from 0 (normal - no symptoms present) to 6 (severely disabled; helpless; complete assistance needed). Higher scores indicate greater disease symptom severity. Negative change from baseline indicates an improvement in the participant's condition.
Time Frame: Baseline, Day 84
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 90 | 93
score on a scale | -0.0 (0.07) | -0.1 (0.07)
Statistical Analysis 1: Comparison: Placebo vs SAGE-718; Test type: Superiority; p = 0.2923, MMRM — The p-value was obtained from MMRM model which includes treatment, visit, treatment-by-visit interaction as categorical covariates, and CGI at baseline as a continuous covariate; Difference in LS Means = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.10 — Difference was calculated as SAGE-718 - placebo

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. A TEAE is defined as an AE with onset after the start of the IP, or any worsening of a pre-existing medical condition/AE with onset after the start of the IP and throughout the study.
Time Frame: Up to last follow-up visit (up to Day 112)
Population: The safety analysis set included all participants who were administered IP.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SAGE-718
Number analyzed (Participants) | 94 | 95
percentage of participants | 75.5 | 62.1

ADVERSE EVENTS:
Time Frame: Up to last follow-up visit (up to Day 112)
Description: The safety analysis set included all participants who were administered IP.
Arm/Group | Placebo | SAGE-718
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/95
Serious Adverse Events (participants affected / at risk) | 6/94 | 3/95
Other Adverse Events (participants affected / at risk) | 29/94 | 18/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | SAGE-718 (N=95)
Fall (Injury, poisoning and procedural complications) | 2 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=94) | SAGE-718 (N=95)
Fall (Injury, poisoning and procedural complications) | 10 | 11
Nausea (Gastrointestinal disorders) | 10 | 2
Irritability (Psychiatric disorders) | 7 | 2
Nasopharyngitis (Infections and infestations) | 6 | 2
Suicidal ideation (Psychiatric disorders) | 5 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2024-08-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT05107128/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT05107128/SAP_001.pdf